CLINICAL TRIAL: NCT04143477
Title: An Open-Label, Single and Multiple Dose Study to Evaluate the Pharmacokinetics and Safety of ASP015K in Healthy Chinese Subjects
Brief Title: A Study to Evaluate the Pharmacokinetics and Safety of ASP015K in Healthy Chinese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma China, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 015K-CL-CNA1
Record Dates: First submitted 2019-10-27; First posted 2019-10-29 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Healthy Volunteers
Keywords: peficitinib; ASP015K; pharmacokinetics
MeSH Terms: interventions — peficitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Peficitinib 50 mg (Experimental): Participants will receive a single dose of 50 milligrams (mg) under fasted condition Day 1, followed by multiple doses of 50 mg under fed condition once daily in the morning from Day 8 till Day 13.
  Interventions: Drug: peficitinib
- Peficitinib 100 mg (Experimental): Participants will receive a single dose of 100 mg under fasted condition Day 1, followed by multiple doses of 100 mg under fed condition once daily in the morning from Day 8 till Day 13.
  Interventions: Drug: peficitinib
- Peficitinib 150 mg (Experimental): Participants will receive a single dose of 150 mg under fasted condition Day 1, followed by multiple doses of 150 mg under fed condition once daily in the morning from Day 8 till Day 13.
  Interventions: Drug: peficitinib

INTERVENTIONS:
Drug: peficitinib — Oral
  Other Names: ASP015K

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics and safety of ASP015K after single-dose and multiple-dose administration in healthy Chinese participants.

ELIGIBILITY:
Inclusion Criteria:

* Normal Body Mass index (BMI) and weight: BMI[= weight kg/(height m)^2] > 19 kg/m^2 and ≤ 24 kg/m^2, the weight is no less than 50 kg for male and 45 kg for female at screening.
* Female subject must either: Be of non-childbearing potential, postmenopausal (defined as at least 1 year without any menses) prior to screening, or documented surgically sterile. Or, if of childbearing potential: agree not to try to become pregnant during the study and for 60 days after the final study drug administration, must have a negative pregnancy at Screening and Day -1, and if heterosexually active, agree to consistently use 1 form of highly effective birth control starting at Screening and throughout the study period, and for 60 days after the final study drug administration.
* Female subject must agree not to breastfeed starting at Screening and throughout the study period, and for 60 days after the final study drug administration.
* Female subject must not donate ova starting at Screening and throughout the study period, and for 60 days after the final study drug administration.
* Male subject and female spouse/partners who are of childbearing potential must be using 1 form of highly effective birth control starting at Screening and throughout the study period, and for 90 days after the final study drug administration.
* Male subject must not donate sperm starting at Screening and throughout the study period, and for 90 days after the final study drug administration.
* Subject agrees not to participate in another interventional study while participating in the present study, defined as signing the informed consent form until completion of the last study visit.

Exclusion Criteria:

* Female subject who has been pregnant within 6 months prior to screening or breast feeding within 3 months prior to screening.
* Subject has a known or suspected hypersensitivity to ASP015K, or any components of the formulation used.
* Subject has any of the liver chemistry tests (aspartate aminotransferase [AST], alanine aminotransferase [ALT], alkaline phosphatase [ALP], gamma-glutamyl transferase [GGT] and total bilirubin [TBL]) above the upper limit of normal on Day -1. In such a case, the assessment may be repeated once.
* Subjects who meet any of the following criterion for laboratory tests on Day -1. Normal ranges of each test specified at the study site or test/assay organization will be used as the normal ranges in this study. In such a case, the assessment may be repeated once.

  * Hematology: a deviation of +20% from the upper limit or -20% from the lower limit of the normal range, and clinically significant.
  * Blood biochemistry: a deviation from the normal range regarding serum creatinine, serum electrolytes (Na, K, and Cl), or fasting blood glucose; a deviation of +20% from the upper limit or -20% from the lower limit of the normal range regarding laboratory test items other than above, and clinically significant. However, the lower limit of the normal range will not be established for lactate dehydrogenase (LD), creatinine kinase (CK), total cholesterol, triglyceride, urea, serum creatinine, and uric acid, whose deviation from the lower limit is considered not clinically significant.
  * Urinalysis: a deviation from the normal range of each urinalysis test item.
* Subject has any clinically significant history of allergic conditions (including drug allergies, asthma, eczema, or anaphylactic reactions, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Subject has any history or evidence of any clinically significant cardiovascular, gastrointestinal endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, respiratory,pulmonary, neurologic, cerebrovascular, lymphatic, dermatologic, psychiatric, renal, and/or other major disease or malignancy.
* Subject has/had febrile illness or symptomatic, viral, bacterial (including upper respiratory infection), or fungal (noncutaneous) infection within 1 week prior to Day -1.
* Subject has any clinically significant abnormality in the physical examination, 12-lead electrocardiogram (ECG) and protocol defined clinical laboratory tests at Screening or Day -1.
* Subject has a pulse rate < 45 or > 100 bpm; systolic blood pressure (SBP) > 140 mmHg; diastolic blood pressure (DBP) > 90 mmHg (measurements taken after subject has been resting in sit position for 5 min; pulse will be measured automatically) at screening or on Day -1. If the pulse rate or blood pressure exceeds the limits above, 1 additional test can be taken.
* Subjects with abnormal body temperature, defined as axillary temperature >37.3 ºC or <35.0 ºC at Screening or Day -1.
* Subject has a corrected QT interval (QTcF) of > 430 ms (for males) and > 450 ms (for females) at screen or on Day -1(at screen and on Day-1, will be performed). If the QTcF exceeds the limits above on Day-1, 1 additional ECG test can be taken.
* Subject has any history or evidence of congenital short QT syndrome(defined as QTc < 330 ms).
* Subject has any history of gastrointestinal resection (excepted appendectomy)..
* Subject has developed upper gastrointestinal symptoms within 1 week prior to Day -1.
* Subject applies to any of the following concerns with regard to tuberculosis.

  * History of active tuberculosis
  * Abnormalities detected in a chest X-ray test at Screening
  * Contact with infectious tuberculous patients
  * T-spot or Quantiferon Gold test show tuberculosisinfection positive.
* Subject applies to any of the following concerns with regard to infection other than tuberculosis.

  * Complication or history of severe herpes zoster or herpes zoster disseminated.
  * At least twice of relapse of localized herpes zoster
  * Inpatient hospital care for severe infectious diseases within 90 days prior to Day -1
  * Treatment with intravenous antibiotics within 90 days prior to Day -1 (prophylactic antibiotics are not applicable).
  * Other than above, with a high risk of developing infectious disease (subjects with urethral catheterisation etc.).
* Subject has vaccination of live vaccines or live attenuated vaccines within 56 days prior to Day -1 (inactivated vaccines such as influenza vaccine and pneumococcal vaccines are not applicable.).
* Subject has used any prescribed or nonprescribed drugs (including vitamins or natural and herbal remedies, e.g. St. John's Wort) in the 2 weeks prior to study drug administration.
* Subject has a history of smoking more than 10 cigarettes (or equivalent amount of tobacco) per day within 3 months prior to admission to the clinical unit.
* Subject has a history of drinking more than 21 units of alcohol per week (1 unit = 10 g pure alcohol = 250 mL of beer [5%] or 35 mL of spirits [35%] or 100 mL of wine [12%]) (> 14units of alcohol for female subjects) within 3 months prior to admission to the clinical unit or the subject tests positive for alcohol or drugs of abuse at Screening or Day -1 (amphetamines,barbiturates, benzodiazepines, cannabinoids, cocaine, and opiates).
* Subject has used any drugs of abuse within 3 months prior to admission to the clinical unit.
* Subject has had significant blood loss, donated 1 unit (450 mL) of blood or more, or received a transfusion of any blood or blood products within 60 days or donated plasma within 7 days prior to Day -1.
* Subject has a positive serology test for hepatitis B surface antigen (HBsAg), antihepatitis A virus (immunodeficiency virus [Ig]M), anti-hepatitis C virus, anti-hepatitis B core or antihuman immunodeficiency virus (HIV) at Screening.
* Subject has participated in any clinical study or has been treated with any investigational drugs within 3 moths prior to screening.
* Subject has any condition which makes the subject unsuitable for study participation.
* Subject is an employee of the Astellas Group, Clinical Research Organization (CRO) or the clinical unit.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2019-12-05 (Actual); Primary Completion 2020-12-21 (Actual); Study Completion 2020-12-21 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | Up to Day 20
  An AE is defined as any untoward medical occurrence in a participant administered a study drug or who has undergone study procedures and which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unintended sign (including an abnormal laboratory finding), symptom or disease temporally associated with the use of a study drug, whether or not related to the study drug.
  An AE is considered "serious" if, in the view of either the investigator or Sponsor, it results in any of the following outcomes: Death, life-threatening, persistent or significant disability/incapacity, congenital anomaly or birth defect, hospitalization, or medically important event.
Number of participants with laboratory value abnormalities and/or AEs | Up to Day 20
  Number of participants with potentially clinically significant laboratory values.
Number of participants with vital sign abnormalities and/or AEs | Up to Day 20
  Number of participants with potentially clinically significant vital sign values.
Number of participants with 12-lead electrocardiogram (ECG) abnormalities and/or AEs | Up to Day 20
  Number of participants with potentially clinically significant 12-ECG values.
Number of participants with physical examination abnormalities and/or AEs | Up to Day 20
  Number of participants with potentially clinically significant physical examination observations.
Pharmacokinetics (PK) of peficitinib: Area under the concentration-time curve (AUC) from the time of dosing extrapolated to time infinity (AUCinf) | On Day 1
  AUCinf will be recorded from the PK serum samples collected.
PK of peficitinib: AUC from the time of dosing to the last measurable concentration (AUClast) | On Day 1 and 8
  AUClast will be recorded from the PK serum samples collected.
PK of peficitinib: AUC from the time of dosing to 24 hours post dose (AUC24h) | On Day 1, 8 and 13
  AUC24h will be recorded from the PK serum samples collected.
PK of peficitinib: Apparent total systemic clearance after extravascular dosing (CL/F) | On Day 1 and 13
  CL/F will be recorded from the PK serum samples collected.
PK of peficitinib: Maximum concertation (Cmax) | On Day 1, 8 and 13
  Cmax will be recorded from the PK serum samples collected.
PK of peficitinib: Terminal elimination rate constant (Lambdaz) | On Day 1 and 13
  Lambdaz will be recorded from the PK serum samples collected.
PK of peficitinib: Terminal elimination half-life (t1/2) | On Day 1 and 13
  t1/2 will be recorded from the PK serum samples collected.
PK of peficitinib: Time of the maximum concentration (tmax) | On Day 1, 8 and 13
  tmax will be recorded from the PK serum samples collected.
PK of peficitinib: Apparent volume of distribution during the terminal elimination phase after single extravascular dosing (VzF) | On Day 1
  VzF will be recorded from the PK serum samples collected.
PK of peficitinib: Concentration immediately prior to dosing at multiple dosing (Ctrough) | On Day 9 to 12 and 13
  Ctrough will be recorded from the PK serum samples collected.
PK of peficitinib: Concentration at 24 hours post dosing (C24h) | On Day 13
  C24h will be recorded from the PK serum samples collected.
PK of peficitinib: Peak trough ratio (PTR) | On Day 13
  PTR will be recorded from the PK serum samples collected.
PK of peficitinib: Accumulation ratio calculated using AUC (Rac(AUC24h)) | On Day 13
  Rac(AUC) will be recorded from the PK serum samples collected.
PK of peficitinib: Accumulation ratio calculated using the maximum concentration (Rac (Cmax)) | On Day 13
  Rac(Cmax)will be recorded from the PK serum samples collected.
PK of peficitinib metabolite: AUCinf | On Day 1
  AUCinf will be recorded from the PK serum samples collected.
PK of peficitinib metabolite: AUClast | On Day 1 and 8
  AUClast will be recorded from the PK serum samples collected.
PK of peficitinib metabolite: AUC24h | On Day 1, 8 and 13
  AUC24h will be recorded from the PK serum samples collected.
PK of peficitinib metabolite: Cmax | On Day 1, 8 and 13
  Cmax will be recorded from the PK serum samples collected.
PK of peficitinib metabolite: Lambdaz | On Day 1 and 13
  Lambdaz will be recorded from the PK serum samples collected.
PK of peficitinib metabolite: t1/2 | On Day 1 and 13
  t1/2 will be recorded from the PK serum samples collected.
PK of peficitinib metabolite: tmax | On Day 1, 8 and 13
  tmax will be recorded from the PK serum samples collected.
PK of peficitinib metabolite: Ctrough | On Day 9 to 12 and 13
  Ctrough will be recorded from the PK serum samples collected.
PK of peficitinib metabolite: C24h | On Day 13
  C24h will be recorded from the PK serum samples collected.
PK of peficitinib metabolite: PTR | On Day 13
  PTR will be recorded from the PK serum samples collected.
PK of peficitinib metabolite: Rac(AUC24h) | On Day 13
  Rac(AUC24h) will be recorded from the PK serum samples collected.
PK of peficitinib metabolite: Rac(Cmax) | On Day 13
  Rac(Cmax) will be recorded from the PK serum samples collected.
PK of peficitinib metabolite: Metabolite to parent ratio of the area under the concentration-time curve corrected by the molecular weight ratio of parent to metabolite (MPR) | On Day 1, 8 and 13
  MPR will be recorded from the PK serum samples collected.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Moniter, Senior Manager, Study Director — Astellas Pharma China, Inc.
Locations (1):
- Site CN86001, Beijing, China

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Derived] Gao X, He X, Oshima H, Miyatake D, Otsuka Y, Kato K, Cai C, Wojtkowski T, Song N, Kaneko Y, Shi A. Pharmacokinetics and Safety of Single and Multiple Doses of Peficitinib (ASP015K) in Healthy Chinese Subjects. Drug Des Devel Ther. 2022 May 9;16:1365-1381. doi: 10.2147/DDDT.S359501. eCollection 2022. PMID 35586186